CLINICAL TRIAL: NCT06360042
Title: Anti-PD-1/PD-L1 Combined With Anti-angiogenic Agents as First-line Therapy for Unresectable Hepatocellular Carcinoma: a Multicenter, Randomized, Open-label Trial
Brief Title: Anti-PD-1/PD-L1 Combined With Anti-angiogenic Agents as First-line Treatment for Unresectable HCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA-HCC-II-021
Record Dates: First submitted 2024-02-27; First posted 2024-04-11 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2023-11

CONDITIONS: Unresectable Hepatocellular Carcinoma
MeSH Terms: interventions — apatinib; Bevacizumab; camrelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1 (Experimental): Adebrelimab（1200mg iv q3w） plus Apatinib(250mg po qd)
  Interventions: Drug: Adebrelimab plus Apatinib
- 2 (Experimental): Adebrelimab（1200mg iv q3w）plus Bevacizumab(15mg/kg iv q3w)
  Interventions: Drug: Adebrelimab plus Bevacizumab
- 3 (Experimental): Camrelizumab (200mg iv q2w) plus Apatinib(250mg po qd)
  Interventions: Drug: Camrelizumab plus Apatinib

INTERVENTIONS:
Drug: Adebrelimab plus Apatinib — Adebrelimab 1200mg intravenously every 3 weeks plus Apatinib 250mg orally once daily
  Arms: 1
Drug: Adebrelimab plus Bevacizumab — Adebrelimab 1200mg intravenously plus Bevacizumab 15 mg/kg intravenously every 3 weeks
  Arms: 2
Drug: Camrelizumab plus Apatinib — camrelizumab 200mg intravenously every 2 weeks plus Apatinib 250mg orally once daily
  Arms: 3

SUMMARY:
This is a multicenter, randomized, open-label clinical study to evaluate the efficacy and safety of Adebrelimab plus Apatinib (cohort 1), or Adebrelimab plus Bevacizumab (cohort 2), or Camrelizumab plus Apatinib (cohort 3) as first-line treatment of unresectable HCC.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic and/or unresectable Hepatocellular Carcinoma (HCC)
* No prior systemic therapy for HCC. Previous use of herbal therapies/traditional Chinese medicines with anti-cancer activity included in the label is allowed.
* BCLC stage B or C, and not suitable for surgical or local therapy, or has progressed following surgical and/or local therapy
* At least one measurable lesion per RECIST v1.1
* ECOG Performance Status of 0 or 1
* Child-Pugh class of A5 to B7
* Adequate organ function

Exclusion Criteria:

* Known hepatocholangiocarcinoma, sarcomatoid HCC, mixed cell carcinoma and lamellar cell carcinoma; other active malignant tumor except HCC within 5 years or simultaneously
* Moderate-to-severe ascites with clinical symptoms
* History of gastrointestinal hemorrhage within 6 months prior to the start of study treatment or clear tendency of gastrointestinal hemorrhage
* Abdominal fistula, gastrointestinal perforation or intraperitoneal abscess within 6 months prior to the start of study treatment
* Known genetic or acquired hemorrhage or thrombotic tendency
* Thrombosis or thromboembolic event within 6 months prior to the start of study treatment
* Hypertension that can not be well controlled through antihypertensive drugs Factors to affect oral administration
* History of hepatic encephalopathy
* Previous or current presence of metastasis to central nervous system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
12-month overall survival rate | Up to approximately 3 years

SECONDARY OUTCOMES:
ORR | Up to approximately 3 years
  Assessed by the investigator per RECIST v1.1 criteria
DCR | Up to approximately 3 years
  Assessed by the investigator per RECIST v1.1 criteria
DoR | Up to approximately 3 years
  Assessed by the investigator per RECIST v1.1 criteria
TTR | Up to approximately 3 years
  Assessed by the investigator per RECIST v1.1 criteria
TTP | Up to approximately 3 years
  Assessed by the investigator per RECIST v1.1 criteria
PFS | Up to approximately 3 years
  Assessed by the investigator per RECIST v1.1 criteria
OS | Up to approximately 3 years
safety according to NCI Common Terminology Criteria for Adverse Events, version 5.0. | Up to approximately 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhou, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No